CLINICAL TRIAL: NCT05612230
Title: A Lifecourse Map of Common Diseases and Rare Diseases in China
Brief Title: A Lifecourse Map of Diseases in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: National Health Medical Data (North Center) (Unknown)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2022-DISEASE
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Common Diseases; Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients: The diseases were included based on the results of the preliminary data exploration and standardization according to ICD-10.
  Interventions: Other: Data analysis

INTERVENTIONS:
Other: Data analysis — Data analysis is based on a single database from the National Health Medical Data (North Center).

SUMMARY:
The purpose of this study is to form a chronological map of common diseases and rare diseases in Chinese population by determining the prevalence of different diseases in each age group.

DETAILED DESCRIPTION:
Studying the distribution of various diseases in specific populations can help explore the causes of diseases, elucidate the distribution patterns, and develop preventive and control measures. Based on an overall assessment of prevalence, the combination of relevant results with age at diagnosis for multiple diseases is important for further understanding of the distribution of diseases at the population level. Therefore, this study aims to form a chronological map of common diseases and rare diseases in Chinese population by determining the prevalence of different diseases in each age group, thus providing a reference for more effective prevention, diagnosis and treatment of diseases.

ELIGIBILITY:
Inclusion Criteria:

1. All inpatients within the period of January 1, 2017 to December 31, 2021.
2. Patients with discharge diagnosis.
3. Patients with accurate gender and age records.

Exclusion Criteria:

1. Morbidity and mortality due to external causes, i.e. injuries, poisonings and other adverse events due to external environment and accidents.
2. Pregnancy-related conditions.
3. Symptoms, signs, abnormal clinical and laboratory findings.
4. Traditional Chinese Medicine diagnosis records.
5. Patients with incorrect or missing disease codes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients within the period of January 1, 2017 to December 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 40000000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
age-specific prevalence rate | between January 1, 2017 and December 31, 2021
  Age-specific prevalence rate stratified by sex were calculated by dividing the number of incident cases with a current disease by the total number of people in the study population during that time period.
sex-specific prevalence rate | between January 1, 2017 and December 31, 2021
  Sex-specific prevalence rate stratified by age for 10-year bands were calculated by dividing the number of incident cases with a current disease by the total number of people in the study population during that time period.

SECONDARY OUTCOMES:
total cost of hospitalization | between January 1, 2017 and December 31, 2021
  Total cost of hospitalization and deductibles for the total population and for each age group of diseases are described by mean (SD) values.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China